CLINICAL TRIAL: NCT02427412
Title: Evaluation of Intraarticular Tranexamic Acid to Reduction of Total Blood Loss Following Knee-Arthroplasty - A Randomized, Prospective, Placebo-Controlled Study
Brief Title: Evaluation of Intraarticular Tranexamic Acid to Reduction of Total Blood Loss Following Knee-Arthroplasty
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hvidovre University Hospital (Other)
Responsible Party: Principal Investigator, Christian Skovgaard Nielsen, MD, Hvidovre University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: H-3-2013-134
Record Dates: First submitted 2015-04-20; First posted 2015-04-28 (Estimated); Last update posted 2015-08-17 (Estimated); Status verified 2015-05

CONDITIONS: Blood Loss; Postoperative Blood Loss; Thromboembolic Complications
Keywords: Tranexamic Acid; Knee Arthroplasty; Blood loss; Blood transfusion; Thrombolic complication; Total blood loss 24 h after ended surgery.; Total blood loss 2 days after ended surgery.
MeSH Terms: conditions — Hemorrhage; Postoperative Hemorrhage | interventions — Tranexamic Acid; Saline Waters

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- IA Tranexamic acid + IV Tranexamic Acid (Active Comparator): 3 gram of Tranexamic acid diluted into 30 ml Saline Water injected into the knee capsula after ended surgery + 1 g of Tranexamic acid injected intravenous at the start of surgery.
  Interventions: Drug: Tranexamic Acid
- IA Saline Water + IV tranexamic Acid (Placebo Comparator): 30 ml Saline Water injected into the knee capsula after ended surgery + 1 g of Tranexamic acid injected intravenous at the start of surgery.
  Interventions: Drug: Saline water; Drug: Tranexamic Acid

INTERVENTIONS:
Drug: Tranexamic Acid — An anti-fibrinolytic drug injected into the knee joint at the end of surgery, 3 g diluted in 30 ml saline water.
  Other Names: Cyclokapron
  Arms: IA Tranexamic acid + IV Tranexamic Acid
Drug: Saline water — 30 ml of Saline water injected into the knee capsula at the end of surgery.
  Other Names: NaCl water
  Arms: IA Saline Water + IV tranexamic Acid
Drug: Tranexamic Acid — An anti-fibrinolytic drug injected intravenous at the beginning of surgery for BOTH groups.
  Other Names: Cyklocapron

SUMMARY:
A randomized, prospective, placebo-controlled study which aims to evaluate the effect of combined intraarticular and intravenous Tranexamic acid on total blood loss following unilateral knee replacement versus only intravenous tranexamic acid.

DETAILED DESCRIPTION:
Intravenous (IV) Tranexamic acid is already well-established and well-documented regarding significant effect on reducing blood loss following knee replacement. A few studies more shown a similar effect of intraarticular (IA) injected Tranexamic acid into the knee joint at the end of surgery for knee replacement.

In this study investigators therefore investigate the possible combined effect of added intraarticular tranexamic acid to conventional intravenous Tranexamic acid.

ELIGIBILITY:
Inclusion Criteria:

* > 18 years old
* Unilateral knee replacement
* Must be able to give oral and written consent

Exclusion Criteria:

* General Anesthetized
* Allergic to Tranexamic acid
* In treatment with the following anticoagulants: Adenosine diphosphate receptor inhibitors or vitamin K antagonist within in the last 5 days. Factor Xa inhibitor and thrombin inhibitor.
* Use of oral anticonceptive.
* Reduced kidney function (S-creatinine > 120 micromol/L)
* Medicine or alcohol abuse
* Females with menstruation within the last 12 mounts.
* Any kind of cancer disease
* Rheumatoid arthritis
* Have participated in a clinical trial within the last 30 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2014-01; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Total estimated blood loss | 24 hours surgery

SECONDARY OUTCOMES:
Total estimated blood loss | 2 days after surgery
Thromboembolic complications | 90 days postoperative
  90 days followup for thromboembolic complications.
Blood transfusion | while hospitalized expected 3 days.
  Estimate the extent of blood transfusions during admission and readmission in relation to the knee replacement

CONTACTS AND LOCATIONS:
Overall Officials: Henrik Husted, PhD, Study Director — Hvidovre University Hospital
Locations (1):
- Hvidovre University Hospital, Hvidovre, Denmark